CLINICAL TRIAL: NCT03211234
Title: A Multi-Center, Randomized, Double Masked and Active Controlled Phase II Study Assessing the Efficacy and Safety of Intravitreal Injections of DE-122 in Combination With Lucentis® Compared to Lucentis® Monotherapy in Subjects With Wet Age-related Macular Degeneration - AVANTE Study
Brief Title: Study Assessing the Efficacy and Safety of Intravitreal Injections of DE-122 in Combination With Lucentis® Compared to Lucentis® Monotherapy in Wet Age-related Macular Degeneration Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36-002
Record Dates: First submitted 2017-07-06; First posted 2017-07-07 (Actual); Results first posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-06

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 2.0 mg DE-122 (Experimental): 2.0 mg DE-122 and Lucentis ® 0.5 mg
  Interventions: Drug: 2.0 mg DE-122 Injectable Solution + Lucentis
- 4.0 mg DE-122 (Experimental): 4.0 mg DE-122 and Lucentis ® 0.5 mg
  Interventions: Drug: 4.0 mg DE-122 Injectable Solution + Lucentis
- Sham (Sham Comparator): Sham and Lucentis ® 0.5 mg
  Interventions: Drug: Lucentis

INTERVENTIONS:
Drug: 2.0 mg DE-122 Injectable Solution + Lucentis — Subjects will receive 6 monthly intravitreal injections of low dose DE-122 in the study eye, in combination with Lucentis.
  Arms: 2.0 mg DE-122
Drug: 4.0 mg DE-122 Injectable Solution + Lucentis — Subjects will receive 6 monthly intravitreal injections of high dose DE-122 in the study eye, in combination with Lucentis.
  Arms: 4.0 mg DE-122
Drug: Lucentis — Subjects will receive 6 monthly intravitreal injections of Sham in the study eye, in combination with Lucentis.
  Arms: Sham

SUMMARY:
To assess the safety and efficacy of repeated intravitreal injections of DE-122 (low dose and high dose) given in combination with Lucentis® in subjects with wet age-related macular degeneration (AMD) compared with Lucentis® alone.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed written informed consent
* Diagnosis of active choroidal neovascularization secondary to wet AMD
* BCVA of 65 to 25 ETDRS letters (20/50 to 20/320) in the study eye
* BCVA of 25 ETDRS letters (20/320) or better in the fellow eye

Exclusion Criteria:

[Ocular]

* Use or anticipated use of any intravitreal, periocular or photodynamic therapy in the study eye for the treatment of AMD within a specified timeframe prior to Visit 1 and throughout the study
* Uncontrolled or advanced glaucoma, chronic hypotony or vitrectomy in the study eye
* Evidence of any other ocular disease other than exudative age-related macular degeneration in the study eye that may confound the outcome of the study
* Need for ocular surgery in the study eye during the course of the study
* Presence or history of certain ocular or periocular pathology or conditions that could limit the ability to perform examinations

[Non-ocular]

* Allergy or hypersensitivity to study drug product, fluorescein dye or other study related procedures and medications
* Current or history of certain systemic conditions, abnormalities or therapies that would render a subject a poor candidate for the study
* Participation in other investigational drug or device clinical trials within 30 days prior to randomization or planning to participate in other investigational drug or device clinical trials for the duration of the study
* Females who are pregnant or lactating and females of child-bearing potential who are not using adequate contraceptive precautions and men who do not agree to practice an acceptable method of contraception throughout the course of the study
* Unable to comply with study procedures or follow-up visits

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (10):
  - Retina Research Institute, Gilbert, Arizona
  - Retina-Vitreous Associates, Beverly Hills, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Colorado Retina Associates, Golden, Colorado
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Retina Reseach Center, Austin, Texas
  - Retina Consultants of Houston, Houston, Texas
  - Valley Retina Insititute, McAllen, Texas
- Philippines (4):
  - Asian Eye Institute, Makati City
  - Peregrine Eye and Laser Institute, Makati City
  - The Medical City, Pasig
  - St. Luke's Medical center Quezon City, Quezon City

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham: Sham and Lucentis
  Lucentis: Subjects will receive 6 monthly intravitreal injections of Sham in the study eye, in combination with Lucentis.
- 2.0 mg DE-122: Low Dose DE-122 and Lucentis
  DE-122 Injectable Solution + Lucentis: Subjects will receive 6 monthly intravitreal injections of low dose DE-122 in the study eye, in combination with Lucentis.
- 4.0 mg DE-122: High Dose DE-122 and Lucentis
  DE-122 Injectable Solution + Lucentis: Subjects will receive 6 monthly intravitreal injections of high dose DE-122 in the study eye, in combination with Lucentis.
Period: Overall Study
Arm/Group | Sham | 2.0 mg DE-122 | 4.0 mg DE-122
Started | 17 | 31 | 28
Completed | 16 | 30 | 25
Not Completed | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham | 2.0 mg DE-122 | 4.0 mg DE-122 | Total
Number analyzed (Participants) | 17 | 31 | 28 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.4 (9.18) | 72.1 (7.34) | 75.6 (9.84) | 74.1 (8.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 15 | 41
  Male | 5 | 17 | 13 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 9 | 9 | 4 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 1 | 0 | 1
  White | 8 | 20 | 24 | 52
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 22 | 25 | 56
  Philippines | 8 | 9 | 3 | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) at Week 24
Description: BCVA is the primary efficacy variable for this study, and mean change from baseline in BCVA at Week 24 is the primary efficacy endpoint.
  An increase in the number of letters read correctly means that vision has improved.The lower the number of letters read correctly on the eye chart, the worse the vision.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Sham | 2.0 mg DE-122 | 4.0 mg DE-122
Number analyzed (Participants) | 17 | 31 | 28
letters | 4.35 (8.937) | 0.87 (11.485) | -1.70 (10.550)

ADVERSE EVENTS:
Time Frame: From Inform consent to the end of the study at week 32.
Arm/Group | Sham | 2.0 mg DE-122 | 4.0 mg DE-122
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/31 | 1/28
Serious Adverse Events (participants affected / at risk) | 1/17 | 1/31 | 4/28
Other Adverse Events (participants affected / at risk) | 5/17 | 10/31 | 10/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sham (N=17) | 2.0 mg DE-122 (N=31) | 4.0 mg DE-122 (N=28)
Cataract (Eye disorders) | 0 | 1 | 0
Subretinal fluid (Eye disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sham (N=17) | 2.0 mg DE-122 (N=31) | 4.0 mg DE-122 (N=28)
Conjunctival hyperaemia (Eye disorders) | 0 | 2 | 4
Eye pain (Eye disorders) | 0 | 4 | 1
Conjunctival haemorrhage (Eye disorders) | 2 | 3 | 0
Conjunctival oedema (Eye disorders) | 0 | 1 | 2
Erythema of eyelid (Eye disorders) | 0 | 1 | 2
Retinal haemorrhage (Eye disorders) | 0 | 3 | 3
Eyelid oedema (Eye disorders) | 0 | 1 | 3
Visual impairment (Eye disorders) | 0 | 1 | 2
Intraocular pressure increased (Investigations) | 0 | 2 | 1
Dry Eye (Eye disorders) | 0 | 2 | 0
Vitreous hemorrhage (Eye disorders) | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 2
Presyncope (Nervous system disorders) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT03211234/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT03211234/SAP_001.pdf